CLINICAL TRIAL: NCT03189810
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Cannabis Use and Cognitive Outcomes in Schizophrenia
Acronym: rTMSCANSZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tony George, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 017-2017
Record Dates: First submitted 2017-05-29; First posted 2017-06-16 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Repetitive Transcranial Magnetic Stimulation (rTMS); Schizophrenia; Cannabis Use Disorder; Cognition
Keywords: Sham Repetitive Transcranial Magnetic Stimulation (rTMS); Schizophrenia; Cannabis Use Disorder; Cognitive Function
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The rTMS technicians, participants, research analysts and investigators involved in the study will be blind to the rTMS treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (20Hz) (Experimental): Active rTMS administered with the MagProX100/R30 stimulator equipped with the B65 active coil for dorsolateral prefrontal cortex (DLPFC) stimulator (MagVenture, Farum, Denmark).The randomization order will be determined by a project scientist from Temerty. While the primary aim of this study is not to treat individuals with cannabis dependence, it is imperative that participants attend weekly study visits in an attempt to achieve end of study (Day 28) cannabis abstinence.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Weekly Counselling Session
- Sham rTMS (Sham Comparator): Sham rTMS administered with the MagProX100/R30 stimulator equipped with the B65 placebo coil for DLPFC stimulator (MagVenture, Farum, Denmark). The randomization order will be determined by a project scientist from Temerty. While the primary aim of this study is not to treat individuals with cannabis dependence, it is imperative that participants attend weekly study visits in an attempt to achieve end of study (Day 28) cannabis abstinence.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Weekly Counselling Session

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — On Day 1, the resting motor threshold (RMT) will be determined according to previous published methods [Cardenas-Morales et al. 2013] and the rTMS will be delivered at an intensity of 90% of the participant's RMT. rTMS will be administered at 20 Hz (25 trains, 30 pulses per train, 30 second intertrain interval).
  Arms: Active rTMS (20Hz)
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — On Day 1, the resting motor threshold (RMT) will be determined according to previous published methods [Cardenas-Morales et al. 2013] and the Sham rTMS will be delivered at an intensity of 90% of the participant's RMT. rTMS will be administered at 20 Hz with the B65 placebo coil (25 trains, 30 pulses per train, 30 second intertrain interval).
  Arms: Sham rTMS
Behavioral: Weekly Counselling Session — In order to support participants in their abstinence plan, individual weekly sessions of supportive counselling will be administered over the course of the study on 1 time per week over 4 weeks (28 days of abstinence).

SUMMARY:
The high prevalence of cannabis and other substance use disorders are a major barrier to recovery in people with schizophrenia. Moreover, schizophrenia patients have significant deficits in cognitive function, which may be exacerbated by cannabis use. Complicating these problems is the lack of evidence-based treatments for co-morbid cannabis use disorders (CUDs) in schizophrenia; there are no established pharmacotherapies. Therefore, this study is investigating the effects of high-frequency (20Hz) repetitive transcranial magnetic stimulation (rTMS) on cannabis use disorder and cognitive function in patients with co-morbid schizophrenia/schizoaffective disorder. The proposed study would be the first randomized, double-blind, sham controlled trial of rTMS in patients with schizophrenia and co-morbid CUD. A total of N=40 schizophrenia smokers with co-morbid cannabis use disorder will be assigned to either active rTMS (N=20) or sham rTMS (N=20) as a treatment regimen of 5X/week treatment for four consecutive weeks. All participants will receive weekly behavioral therapy for 4 weeks. The investigators predict that active rTMS will be well-tolerated and superior to sham rTMS for the treatment of CUD in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Male (80%) or Female (20%);
2. Age 18-55;
3. Meet the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for Schizophrenia (SZ) or schizoaffective disorder and cannabis use disorder with physiological dependence;
4. Full scale intelligence quotient (IQ) ≥ 80 determined through the Wechsler Test of Adult Reading (WTAR);
5. Non-smokers OR cigarette smokers as confirmed with Fragerstrom Test for Nicotine Dependence (FTND) score of 5 or higher, self reported smoking of at lest 5 cigarettes per day (measured by the Timeline Follow Back), and verified by a Smokerlyzer test, cut-off as 10 ppm.

Exclusion Criteria:

1. DSM-5 diagnoses of alcohol, substance or polyuse substance use disorder in the past 6 months (other than cannabis/caffeine or nicotine);
2. Currently active suicidal ideation or self-harm (suicidal or non-suicidal) as assessed by the Structured Clinical Interview for DSM-5 (SCID-5);
3. Head injury resulting in loss of consciousness (>5 minutes) and hospitalization;
4. Major neurological or medical illness including seizure disorder or syncope;
5. Metallic implants;
6. History of rTMS treatment;
7. Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The effects of active versus sham rTMS directed to DLPFC on cannabis abstinence in cannabis-dependent patients with schizophrenia as assessed by urine screens for changes in Tetrahydrocannabinol (THC) content. | Weekly (Day 0, Day 7, Day 14, Day 21, Day 28) and at 8 weeks (Follow-up Day 56)
  Urine samples will be collected weekly during the abstinence period and tested by study personnel using the Semi-Quantitative THC Pre-Dosage Test (NarcoCheck®, Villejuif, France).
The effects of active versus sham rTMS directed to DLPFC on cannabis abstinence in cannabis-dependent patients with schizophrenia as assessed by urine screens for changes in Tetrahydrocannabinol (THC) content. | Up to 4 weeks (Day 28) and 8 weeks (Follow-Up Day 56)
  Urine samples at Day 28 and Follow-Up (Day 56) will be sent to CAMH's clinical laboratory for gas chromatography/mass spectrometry (GC/MS) analysis to obtain quantitative THC-COOH and creatinine concentrations. Thus abstinence will also be assessed with combined quantitative urinalysis (<50 ng/ml) and TLFB assessment.

SECONDARY OUTCOMES:
The effects of active (20 Hz) versus sham rTMS on change in cognitive function in cannabis dependent patients with schizophrenia as assessed by a cognitive battery administered at Baseline and at Day 28. | Up to 4 weeks (Day 28) and 8 weeks (Follow-Up Day 56)
  The cognitive battery (Day 28) will include the primary outcome of verbal memory (assessed by HVLT) and will be compared to baseline (Day 1) performance. Cortical inhibition will also be assessed and compared between Day 1 and Day 28 performance.

OTHER OUTCOMES:
The effects of active (20 Hz) versus sham rTMS on change in cannabis craving in cannabis-dependent patients with schizophrenia as assessed by the Marijuana Craving Questionnaire (MCQ). | Up to 4 weeks (Day 28) and 8 weeks (Follow-Up Day 56)
  MCQ will be assessed over time, specifically at Day 1 compared to Day 28.
The effects of active (20 Hz) versus sham rTMS on change in cannabis withdrawal in cannabis-dependent patients with schizophrenia as assessed by the Marijuana Withdrawal Checklist (MWC). | Up to 4 weeks (Day 28) and 8 weeks (Follow-Up Day 56)
  MWC will be assessed over time, specifically at Day 1 compared to Day 28.
The effects of active (20 Hz) versus sham rTMS on psychotic symptoms in cannabis-dependent patients with schizophrenia as assessed by the Calgary Depression Scale for Schizophrenia (CDSS). | Up to 4 weeks (Day 28) and 8 weeks (Follow-Up Day 56)
  CDSS scores will be compared over time, specifically Day 1 compared to Day 28. The depressive subscales within the PANSS will also be compared with the CDSS final score.
The effects of active (20 Hz) versus sham rTMS on psychotic symptoms in cannabis-dependent patients with schizophrenia as assessed by the Positive and Negative Syndrome Scale (PANSS). | Up to 4 weeks (Day 28) and 8 weeks (Follow-Up Day 56)
  PANSS will be compared over time, specifically Day 1 compared to Day 28. The depressive subscales within the PANSS will also be compared with the CDSS final score.

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, MD, FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnstone S, Sorkhou M, Zhang M, Dermody SS, Rabin RA, George TP. Cannabis cravings predict cigarette use in schizophrenia: a secondary analysis from two cannabis abstinence studies. Am J Drug Alcohol Abuse. 2024 Jan 2;50(1):95-105. doi: 10.1080/00952990.2023.2292010. Epub 2024 Jan 12. PMID 38214479
- [Derived] Johnstone S, Lowe DJE, Kozak-Bidzinski K, Sanches M, Castle DJ, Rabin JS, Rabin RA, George TP. Neurocognitive moderation of repetitive transcranial magnetic stimulation (rTMS) effects on cannabis use in schizophrenia: a preliminary analysis. Schizophrenia (Heidelb). 2022 Nov 17;8(1):99. doi: 10.1038/s41537-022-00303-2. PMID 36384966